CLINICAL TRIAL: NCT01297868
Title: Impact of Exercise on Retinal Microvascular Regulation Measured by Dynamic Vessel Analysis in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Other Study IDs: DVAAug-1
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Middle-aged Subjects; Age Range Was 18 to 31 Years; Caucasian Whites; Males and Females
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- exercise group
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise

SUMMARY:
Objective The investigators assessed the acute impact of physical exercise on retinal vessel regulation. This might be of clinical importance if retinal vessel regulation is examined with the very sensitive method of the dynamic vessel analyzer Design Forty middle aged (age range 18 to 31 years, mean age 24 years) healthy subjects (26 female / 14 male) had retinal examinations with static and dynamic vessel analysis prior and after (0.5h, 1.5h, 2.5h) intense exercise of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy middle-aged subjects

Exclusion Criteria:

* volunteers with systemic or ocular diseases

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: healthy middle-aged subjects, unselected volunteers
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
retinal vessel diameter

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Greifswald, Germany